CLINICAL TRIAL: NCT05624229
Title: Efficacy of Proton Pump Inhibitors in Cirrhotic Patients With Acute Variceal Bleeding
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPI-AVB
Record Dates: First submitted 2022-11-12; First posted 2022-11-22 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Upper Gastrointestinal Hemorrhage
Keywords: Proton Pump Inhibitors; Acute Variceal Bleeding; Liver Cirrhosis; Endoscopic Variceal Ligation
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Liver Cirrhosis | interventions — Proton Pump Inhibitors; Omeprazole; Esomeprazole; Rabeprazole; Pantoprazole; ilaprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard group (Placebo Comparator): Early treatment is mainly aimed at correcting hypovolemic shock, preventing gastrointestinal bleeding-related complications, effective control of bleeding, monitoring vital signs and urine output.
  Medical treatment included initiation and maintenance of vasoactive agents as soon as possible for 2 to 5 days, and prophylactic antibiotics (preferably ceftriaxone sodium or quinolones) by intravenous infusion for 5 days.
  Endoscopic intervention was performed within 12 hours after presentation and generally no longer than 24 hours. PPI was stopped immediately after endoscopic treatment.
  Early TIPS is determined according to the technology and concept of each unit.
  Interventions: Drug: No Proton Pump Inhibitors
- Standard group+PPI (Experimental): PPI continued after endoscopic treatment for 5 days.
  Interventions: Drug: Proton Pump Inhibitors

INTERVENTIONS:
Drug: Proton Pump Inhibitors — PPI infusion continued to use for 5 days in experimental group
  Other Names: Drug: Omeprazole; Drug: Esomeprazole; Drug: Rabeprazole; Drug: Pantoprazole; Drug: Ilaprazole; Drug: Lansoprazole
  Arms: Standard group+PPI
Drug: No Proton Pump Inhibitors — PPI infusion stopped in standard group after endoscopy.
  Arms: Standard group

SUMMARY:
Acute Variceal Bleeding (AVB) in patients with liver cirrhosis is a common clinical critical disease. There is little evidence for the effect of proton pump inhibitor (PPI) use in patients with AVB, and there is no study on the efficacy of PPI combined with standard therapy in patients with AVB.

DETAILED DESCRIPTION:
AVB in patients with liver cirrhosis is a common clinical critical disease, with a 6-week mortality rate as high as 20%. Currently, many guidelines recommend the use of vasoactive drugs (terlipressin, somatostatin or octreotide) combined with endoscopic therapy (Endoscopic Variceal Ligation (EVL), endoscopic injection sclerotherapy (EIS) and the use of prophylactic antibiotics for patients with AVB.

PPI is a commonly used antacid agent, which has a significant antacid effect, protects the gastrointestinal mucosa, promotes blood coagulation, healing ulcers, effectively stops bleeding and prevents rebleeding. There is a consensus that PPI should be used before and after endoscopic therapy in patients with non-variceal acute bleeding. However, studies on the efficacy of PPI after EVL are still limited and lack of sufficient convincing. In a randomized controlled study, pantoprazole treatment was found to be associated with significantly smaller ulcers 10 days after elective EVL in secondary prevention patients with cirrhosis. Another randomized controlled study in 2013 found that patients with cirrhosis and AVB treated with PPI for 19 days after endoscopic hemostasis had smaller ulcers and fewer overall side-effects, but there was no statistically significant difference in rate of 5-day treatment failure, 6-week rebleeding rate and 6-week mortality. In 2017, a study included 637 patients with acute bleeding from liver cirrhosis, 80% of whom were treated with acid suppression therapy, and the study found that acid suppression therapy had no significant effect on long-term bleeding rate and mortality. However, negative effects of PPI have been reported in patients with cirrhosis, such as spontaneous bacterial peritonitis and hepatic encephalopathy. It is found that patients with cirrhosis and ascites had an increased risk of first hepatic encephalopathy with PPI use, and also found that patients with cirrhosis had an increased risk of hepatic encephalopathy and death with PPI use. Therefore, PPI use in patients with cirrhosis should be more cautious. However, the duration of PPI use in these studies was long, and there are no data to clarify the effect of short-term PPI use.

At present, there is no consensus among the major guidelines on the use of PPI in patients with acute AVB in liver cirrhosis, and the UK guidelines do not recommend the use of PPI unless accompanied by gastrointestinal ulcer. The use of PPI was not mentioned in the guidelines of the American Endoscopic Society and the European Endoscopic Society. The 2021 Baveno 7 guideline clearly proposes that PPI should be stopped immediately once AVB is identified as cirrhosis. The latest meta-analysis in 2022 showed that the use of PPI before endoscopy may reduce the need for endoscopic hemostasis in patients with upper gastrointestinal tract, but there was no sufficient evidence to confirm the effect on clinical outcomes including 30-day mortality and rebleeding. It can be concluded that there is no consensus on the use of PPI in patients with AVB in cirrhosis, and the recommendations of guidelines lack high-quality studies to improve the convincing.

In summary, there is little evidence for the effect of PPI use in patients with AVB in liver cirrhosis, and there is no study on the efficacy of PPI combined with endoscopic therapy in patients with AVB in liver cirrhosis. Therefore, the investigators planned to design a multicenter prospective randomized controlled trial to explore the efficacy of PPI in cirrhotic patients with AVB. In this study, the following questions were investigated: 1. Can PPI reduce the 5-day treatment failure rate in cirrhotic patients with AVB; 2. Can it reduce the 6-week rebleeding rate, mortality, and complications in patients with liver cirrhosis and AVB.

ELIGIBILITY:
Inclusion Criteria:

1. Liver cirrhosis.
2. The etiology of portal hypertension is cirrhosis.
3. Patients presenting with acute esophageal variceal bleeding proven by emergency endoscopy within 24 hours.
4. Be willing to participate in this clinical study, comply with the study requirements and sign the informed consent

Exclusion Criteria:

1. non-cirrhotic portal hypertension
2. the time from admission to endoscopy was more than 24 hours
3. patients with peptic ulcer or gastroesophageal reflux disease requiring PPI therapy
4. PPI use for more than 2 weeks before admission
5. received endoscopic or interventional therapy within the previous 4 weeks
6. PPI allergy
7. Chronic renal insufficiency (CKD stage 3-5)
8. Severe cardiopulmonary dysfunction (such as heart failure grade 3-4, respiratory failure, etc.)
9. Hepatocellular carcinoma (Barcelona Clinic Liver Cancer (BCLC) stage C and D)
10. other advanced malignancies (life expectancy less than 6 months)
11. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 672 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
5-day treatment failure rate | 5 days
  Failure of initial hemostasis Initial hemostasis was defined as not achieving a 24h bleeding-free period within the first 48h after treatment together with stable vital signs based on Baveno consensus criteria.
  UGI bleeding occurred after initial hemostasis and within 5 days after enrollment was defined as early rebleeding. UGI bleeding was proven to be from esophageal varices.

SECONDARY OUTCOMES:
Rebleeding rate within 42 days | 42 days
  Rebleeding rate within 42 days
Mortality rate within 42 days | 42 days
  Mortality rate within 42 days
Rescure treatment | 42 days
  Number of participants who need of TIPs, re-endoscopy, surgery, etc
Compilcations | 42 days
  Occurrence of chest pain, reflux, nausea, vomiting, dysphagia, ulcer perforation, diarrhea, abdominal pain, headache, hepatic encephalopathy, spontaneous peritonitis, etc